CLINICAL TRIAL: NCT02945254
Title: Effect of Continuous Background Noise at Specific Frequencies on Objective and Subjective Sleep Quality
Brief Title: Effect of Background Noise on Sleep Quality
Acronym: Noise
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, MD, PhD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000982
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Sleep Onset Insomnia
Keywords: sleep onset latency; sleep quality; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Background noise (Active Comparator): Overnight sleep study with filtered white noise
  Interventions: Device: NIghtingale (R) device for filtered white noise (Cambridge Sound Management, Waltham, MA)
- Silence (No Intervention): Overnight sleep study with normal environmental noise

INTERVENTIONS:
Device: NIghtingale (R) device for filtered white noise (Cambridge Sound Management, Waltham, MA)
  Arms: Background noise

SUMMARY:
Insufficient and low-quality sleep is a major public health problem that has been linked to motor vehicle crashes, industrial disasters, and medical and other occupational errors. Persons experiencing sleep insufficiency are also more likely to suffer from chronic diseases such as hypertension, diabetes, depression, and obesity, as well as from cancer, increased mortality, and reduced quality of life and productivity.

The number of people using sleep-inducing drugs to increase or improve sleep is steadily increasing in the last few decades; however, the side effects of these therapies often outweigh the benefits.

A few small trials and anecdotal findings suggest that continuous background (pink or white) noise overnight can improve sleep quality, increase acoustic arousal threshold, and reduce sleep onset latency.

In an attempt to find new, alternative solutions to increase sleep quality in people suffering from insomnia, the investigators would like to test the effect of surrounding filtered white noise on sleep onset latency and subjective sleep quality in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 60

Exclusion Criteria:

* Any sleep disorder
* Use of hypnotics

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Background Noise First, Silence Second: Overnight sleep study with filtered white noise (Nightingale (R) device, Cambridge Sound Management, Waltham, MA) on the first study night, then a 1-week non-treatment period, then Overnight sleep study with normal environmental noise
- Silence First, Background Noise Second: Overnight sleep study with normal environmental noise, then a 1-week non-treatment period, then an Overnight sleep study with filtered white noise (Nightingale (R), Cambridge Sound Management, Waltham, MA)
Period: Overall Study
Arm/Group | Background Noise First, Silence Second | Silence First, Background Noise Second
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Background Noise First, Silence Second | Silence First, Background Noise Second | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (9.1) | 31.6 (10.4) | 30.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency (Mins)
Description: time from lights out to the first epoch of stage 2 NREM sleep
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Background Noise: Overnight sleep study with filtered white noise (NIghtingale (R) Cambridge Sound Management, Waltham, MA)
Arm/Group | Background Noise | Silence
Number analyzed (Participants) | 18 | 18
minutes | 13 [5 to 31] | 19 [12 to 28]
Statistical Analysis 1: Comparison: Background Noise vs Silence; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney) — P<0.05 considered statistically significant

2. Secondary Outcome: Subjective Sleep Quality (VAS)
Description: subjective sleep quality was assessed in the morning with a visual analog scale (VAS) ranging from 1 (worse quality) to 10 (best quality)
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Background Noise | Silence
Number analyzed (Participants) | 18 | 18
units on a scale | 7 [4.7 to 7.3] | 7 [6.8 to 8.3]
Statistical Analysis 1: Comparison: Background Noise vs Silence; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney) — P<0.05 considered statistically significant

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Background Noise | Silence
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02945254/Prot_SAP_ICF_000.pdf